CLINICAL TRIAL: NCT05084755
Title: VAXZEVRIA Intramuscular Injection Specific Use Result Study for the Subjects With Underlying Disease at High-risk for Worsening COVID-19
Brief Title: VAXZEVRIA Japan Post-Marketing Surveillance (PMS) for the Subjects With Underlying Disease at High-risk for Worsening COVID-19
Status: Terminated | Type: Observational
Why Stopped: In Japan, the government purchases VAXZEVRIA and distributes it to medical institutions. Based on Japan VAXZEVRIA vaccination plan, the last vaccination day was Sep. 30, 2022. So it was difficult to continue this study.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8111C00006
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Prevention of Infectious Disease Caused by SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
To provide more information on safety profile of VAXZEVRIA in Japanese subjects, specific drug use result study in subjects with underling disease at higher risk of worsening COVID-19 is planned as an additional pharmacovigilance plan.

The present study aims to collect information on adverse drug reactions or COVID-19 infection after VAXZEVRIA vaccination and to evaluate the safety of this vaccine.

DETAILED DESCRIPTION:
To provide more information on safety profile of VAXZEVRIA in Japanese subjects, specific drug use result study in subjects with underling disease at higher risk of worsening COVID-19 is planned as an additional pharmacovigilance plan.

The present study aims to collect information on adverse drug reactions (local/systemic reactions), adverse events (including Shock/ Anaphylaxis, Thrombosis in combination with thrombocytopenia, Immune-mediated neurological conditions ,Vaccine-associated enhanced disease(VAED) including Vaccine-associated enhanced respiratory disease(VAERD) and Thrombosis) or COVID-19 infection after VAXZEVRIA vaccination and to evaluate the safety of this vaccine

ELIGIBILITY:
Inclusion Criteria:

1. The subjects with underlying disease at high-risk for worsening COVID-19.
2. The adults (in the case of a minor aged less than 20 years, the parent or the legal guardian) who are able to enter their symptoms in the health observation diary and who have been fully informed and have given written consent to the use of the needed information to be part of the observational study.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects with underlying disease at high-risk for worsening COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions, its incidence (%) (number of adverse drug reaction/number of eligible safety analysis population) will be calculated by preferred term (PT). | from the first vaccination date to 28 days after the second vaccination date
  Adverse events that the investigator could not deny the causal relationship with VAXZEVRIA will be treated as adverse drug reactions. Number of adverse drug reactions, its incidence (%) (number of adverse drug reaction/number of eligible safety analysis population) will be calculated by preferred term (PT).
Number of local/systemic reactions and its incidence (%) will be calculated for each reaction and also by grade. Ad hoc analysis might be performed as necessary. | each vaccination day (Day 1) to Day 8
  Local/systemic reactions recorded in health observation diary by subjects and entered by the investigator in eCRF will be treated as specific adverse events and number of local/systemic reactions and its incidence (%) will be calculated for each reaction and also by grade. Ad hoc analysis might be performed as necessary.
Number of the subjects considered to be severe case of COVID-19 and its incidence (%) will be calculated. The subject who required a hospitalization in intensive care unit or use of respirator will be defined as a severe case. | from the first vaccination date to 28 days after the second vaccination date
  Number of the subjects considered to be severe case of COVID-19 and its incidence (%) will be calculated. The subject who required a hospitalization in intensive care unit or use of respirator will be defined as a severe case based on the severity classification reference of "A guide for front-line healthcare workers (MHLW, 2020)". Ad hoc analysis might be performed as necessary.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Research Site, Akita
  - Research Site, Ibaraki
  - Research Site, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home